CLINICAL TRIAL: NCT05995080
Title: The Effectiveness of Chlorhexidine Gluconate Bathing on Prevention of Catheter-Related Bloodstream Infections in Pediatric Intensive Care Unit
Brief Title: The Effectiveness of Chlorhexidine Gluconate on Prevention of Catheter-Related Bloodstream Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Saime Hacer Ozdemir, Principle Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0009-0009-3168-4445
Record Dates: First submitted 2023-07-12; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Central Venous Catheter Related Bloodstream Infection; Catheter-Related Infections; Bloodstream Infection Due to Central Venous Catheter
Keywords: chlorhexidine gluconate; catheter-related bloodstream infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Intervention Model Description: The control and study groups were determined by applying randomization at a ratio of 1:1 to the patients which participated to the study.
Who Masked: Investigator
Masking Description: The control and study groups were determined by applying randomization at a ratio of 1:1 to the patients which participated to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chlorhexidine bathing group (Experimental): Patients aged between 2 months and 18 years with temporary central venous catheter in the pediatric intensive care unit were recruited. Patients younger than 2 months of age, patients with a catheter use of less than 48 hours, patients with a history of allergic reaction with chlorhexidine, patients with a skin condition that interferes with skin cleansing with chlorhexidine, and immunocompromised patients were excluded from the study. Participants of the study were randomized with a ratio of 1:1. In study group, standard bathing will be applied on the first day of insertion of the central venous catheter, and in addition to that it is planned to clean the skin of the patient daily with cleaning pads impregnated with 2% Chlorhexidine gluconate.
  Interventions: Other: clorhexidine gluconate bathing
- standart bathing group (No Intervention): Patients who are included in the study but not intervention group will be treated with standard bathing, which applied in every 72 hours in our facility.

INTERVENTIONS:
Other: clorhexidine gluconate bathing — daily skin cleansing with chlorhexidine gluconate
  Other Names: cathater care practices
  Arms: chlorhexidine bathing group

SUMMARY:
Catheter-related bloodstream infections are associated with increased mortality, morbidity, and length of hospital stay. The incidence has decreased significantly with the strict implementation of preventive bundle cares and checklists in intensive care units. Bathing with solutions containing chlorhexidine has been included in preventive strategies in recent years. Although some studies have shown that chlorhexidine bathing reduces the frequency of hospital-associated infections, there are important differences in management of practice and adherence to practice in different facilities. The majority of the studies conducted include adult patients. According to the CDC guidelines, chlorhexidine bathing is recommended for children over 2 months of age to prevent catheter-related bloodstream infection. The aim of this study is to investigate the effect of daily bathing with 2% chlorhexidine gluconate solution in preventing catheter-related bloodstream infections in pediatric patients with temporary central venous catheters.

DETAILED DESCRIPTION:
In patients with a central catheter for longer than 48 hours, the diagnosis of bloodstream infection will be recorded as laboratory-confirmed bloodstream infections according to CDC diagnostic criteria. Microorganisms detected in cultures will be classified as gram-positive and gram-negative or fungal agents. Infection with the resistant microorganism will be compared with the control group. Catheter colonization; be defined as bacterial growth of more than 15 colonies in the semiquantitative culture or 1000 colonies in the quantitative culture of the catheter segment or hub without clinical symptoms.

Patients in both groups with a central catheter for longer than 48 hours will be treated with a standard bath every 72 hours. In addition to the control group, patients in the study group will be treated daily with 2% chlorhexidine gluconate, and the patients in these two groups will be compared in terms of catheter-related bloodstream infections and catheter colonization.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 2 months and 18 years who had a temporary central venous catheter
* Patients whose follow-up is continued for at least 48 hours with a central venous catheter

Exclusion Criteria:

* Patients younger than 2 months of age
* Patients with a intensive care unit stay shorter than 48 hours
* Immunosuppressive patients
* Patients with a history of allergic reaction to chlorhexidine
* Patients with skin lesions that interfere with skin cleansing with chlorhexidine
* Patients whose family did not give consent

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Catheter-related blood stream infection rates | 2 years.
  In patients with a central catheter for longer than 48 hours, the diagnosis of bloodstream infection will be recorded as laboratory-confirmed bloodstream infections according to CDC diagnostic criteria.
  Microorganisms detected in cultures will be classified as gram-positive and gram-negative or fungal agents. Infection with the resistant microorganism will be compared with the control group.
Catheter colonization rates | 2 years.
  Catheter colonization; be defined as bacterial growth of more than 15 colonies in the semiquantitative culture or 1000 colonies in the quantitative culture of the catheter segment or hub without clinical symptoms.
Demographic features of participants | 2 years.
  The investigators will be evaluating the features below:
  * Age of the patients (months)
  * Sex of patients
  * Weight of patients (kilograms)
  * Height of patiens (centimeters)
Comorbidities of participants | 2 years.
  The investigators will be evaluating the comorbidities in each groups, in order to determine if any of these conditions would interfere with infection rates.
Catheter site of placement | 2 years.
  It will be classified as; femoral, internal jugular, subclavian.
The duration of intensive care unit stay for each participants | 2 years.
  It will be evaluated as days.
Duration of catheter usage | 2 years.
  It will be evaluated as the total amount of time as days.
Number of catheter lumens | 2 years.
  It will be evaluated wether it has 2 or 3 lumens.
Time when catheter is started the use | 2 years.
  It will be noted that the time of intensive care hospitalization that catheter usage started.
  It will be evaluated as days.
Number of catheter dressing changes | 2 years.
  It will be evaluated that the amount of planned or unplanned changes of catheter dressing.
Reason for the catheter removal | 2 years.
  It will be classified as for example; infection, dysfunction, lack of need...
The reason of intensive care hospitalization for each participants | 2 years.
  It will be evaluated that the primary reason that cause for patient to need for intensive care.
PRISM (pediatric risk of mortality) score of the participants | 2 years.
  The Pediatric Risk of Mortality (PRISM) score was developed from the Physiologic Stability Index (PSI) to reduce the number of physiologic variables required for pediatric ICU (PICU) mortality risk assessment and to obtain an objective weighting of the remaining variables.
Need for invasive mechanical ventilation support | 2 years.
  It will be evaluated if the patient needed for invasive mechanical ventilation support or not. If so, how many days is it required will be noted.
Need for hemodialysis catheter usage | 2 years.
  It will be noted that wether the patient has hemodialysis catheter or not.
Presence of parenteral steroid use | 2 years.
  It will be noted that if during the intensive unit care, wether patient need pulse steroid treatment (30milligram/kilogram/day for 3 or more days) or treatment with Prednisolone 2 milligram/kilogram/day or more for 14 or more days

SECONDARY OUTCOMES:
Rate of catheter-related bloodstream infection in patients bathing with 2% chlorhexidine gluconate daily. | Through study completion, 2 years.
  Incidence will be determined by dividing the number of patients who had catheter-related bloodstream infections in patients who underwent daily skin cleansing with chlorhexidine, compared to the total number of patients who underwent daily skin cleansing with chlorhexidine.
  Patients who were treated with a standard bath and those treated with a chlorhexidine bath will be compared.
Rate of catheter colonization in patients bathing with 2% chlorhexidine gluconate daily. | 2 years.
  Incidence will be determined by dividing the number of patients who had catheter colonization in patients who underwent daily skin cleansing with chlorhexidine, compared to the total number of patients who underwent daily skin cleansing with chlorhexidine.
  Patients who were treated with a standard bath and those treated with a chlorhexidine bath will be compared.
Microorganisms that grown in cultures of catheter-related bloodstream infection in patients bathing with 2% chlorhexidine gluconate daily. | 2 years.
  It will be noted which microorganisms grown in the cultures. By classifying microorganisms grown in culture (gram positive, gram negative, fungal infections, etc.), a comparison will be made between the two groups in terms of incidence.
Microorganisms that cause catheter colonization in patients bathing with 2% chlorhexidine gluconate daily. | 2 years.
  It will also be noted which microorganisms grown in the cultures. By classifying microorganisms grown in culture (gram positive, gram negative, fungal infections, etc.), a comparison will be made between the two groups in terms of incidence.
Rate of catheter-related bloodstream infection in patients who applied standard bathing | 2 years
  Incidence will be determined by dividing the number of patients who had catheter-related bloodstream infection in patients who underwent standard bathing to the total number of patients who underwent standard bathing.
  Patients who were treated with a standard bath and those treated with a chlorhexidine bath will be compared.
Rate of catheter colonizsation in patients who applied standard bathing | 2 years
  Incidence will be determined by dividing the number of patients who had catheter colonization in patients who underwent standard bathing to the total number of patients who underwent standard bathing.
  Patients who were treated with a standard bath and those treated with a chlorhexidine bath will be compared.
Microorganisms that grown in cultures of catheter-related bloodstream infection in patients which applied standard bathing | 2 years.
  It will also be noted which microorganisms grown in the cultures. By classifying microorganisms grown in culture (gram positive, gram negative, fungal infections, etc.), a comparison will be made between the two groups in terms of incidence.
Microorganisms that cause catheter colonization in patients which applied standard bathing | 2 years.
  It will also be noted which microorganisms grown in the cultures. By classifying microorganisms grown in culture (gram positive, gram negative, fungal infections, etc.), a comparison will be made between the two groups in terms of incidence.

CONTACTS AND LOCATIONS:
Locations (1):
- IMU, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zerr DM, Milstone AM, Dvorak CC, Adler AL, Chen L, Villaluna D, Dang H, Qin X, Addetia A, Yu LC, Conway Keller M, Esbenshade AJ, August KJ, Fisher BT, Sung L. Chlorhexidine gluconate bathing in children with cancer or those undergoing hematopoietic stem cell transplantation: A double-blinded randomized controlled trial from the Children's Oncology Group. Cancer. 2021 Jan 1;127(1):56-66. doi: 10.1002/cncr.33271. Epub 2020 Oct 20. PMID 33079403
- [Result] Tien KL, Sheng WH, Shieh SC, Hung YP, Tien HF, Chen YH, Chien LJ, Wang JT, Fang CT, Chen YC. Chlorhexidine Bathing to Prevent Central Line-Associated Bloodstream Infections in Hematology Units: A Prospective, Controlled Cohort Study. Clin Infect Dis. 2020 Jul 27;71(3):556-563. doi: 10.1093/cid/ciz874. PMID 31504341